CLINICAL TRIAL: NCT07372014
Title: A Comparative Analysis of the Effectiveness of Nepafenac Combined With a Lubricant Versus a Lubricant Alone in the Treatment of Epiphora Associated With Lacrimal Punctum Stenosis in Mexican Adults
Brief Title: A Comparative Analysis of the Effectiveness of Nepafenac Combined With a Lubricant Versus a Lubricant Alone in the Treatment of Epiphora Associated With Lacrimal Punctum Stenosis
Acronym: CAENLVLTELPMA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEI-2025/09/01
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Epiphora; Punctal Stenosis
Keywords: Lacrimal Apparatus Diseases; Stenosis; Anti-Inflammatory Agents, Non-Steroidal
MeSH Terms: conditions — Lacrimal Apparatus Diseases; Constriction, Pathologic | interventions — nepafenac; Lubricants

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized clinical trial with a follow-up period of two months. Participants will be allocated into two groups through balanced block randomization.
  The first group will receive nepafenac ophthalmic suspension 0.1% once daily, in conjunction with sodium carboxymethylcellulose 0.5% three times daily, over an eight-week period. The second group will be administered a placebo alongside sodium carboxymethylcellulose 0.5% three times daily for the same duration. All assessments will be conducted by a single ophthalmologist.
  Prior to the initiation of treatment, at 4 and 8 weeks into the treatment, a clinical evaluation using a slit lamp will be performed to assess the visibility of the lacrimal punctum, utilizing the Kashkouli scale, and to evaluate epiphora according to the Munk scale. Additionally, baseline measurements of the external diameter and depth of the lacrimal punctum will be obtained using OCT-SA.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Nepafenac 0.1% ophthalmic suspension and lubricant (Experimental): The study participants will be randomly assigned to two groups: the first group will receive treatment with nepafenac 0.1% ophthalmic suspension once daily and sodium carboxymethylcellulose 0.5% (lubricant) three times daily for eight weeks; the second group will receive treatment with placebo and lubricant only, administered three times daily for eight weeks
  Interventions: Drug: Nepafenac and lubricant
- Group 2: placebo and lubricant (Placebo Comparator): The study participants will be randomly assigned to two groups: the first group will receive treatment with nepafenac 0.1% ophthalmic suspension once daily and sodium carboxymethylcellulose 0.5% (lubricant) three times daily for eight weeks; the second group will receive treatment with placebo and lubricant only, administered three times daily for eight weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nepafenac and lubricant — A two-month follow-up will be conducted. The study participants will be randomly assigned to two groups: the first group will receive treatment with nepafenac 0.1% ophthalmic suspension once daily and sodium carboxymethylcellulose 0.5% (lubricant) three times daily for eight weeks; the second group will receive treatment with placebo and lubricant only, administered three times daily for eight weeks
  Arms: Group 1: Nepafenac 0.1% ophthalmic suspension and lubricant
Drug: Placebo — A two-month follow-up will be conducted. The study participants will be randomly assigned to two groups: the first group will receive treatment with nepafenac 0.1% ophthalmic suspension once daily and sodium carboxymethylcellulose 0.5% (lubricant) three times daily for eight weeks; the second group will receive treatment with placebo and lubricant only, administered three times daily for eight weeks
  Arms: Group 2: placebo and lubricant

SUMMARY:
Establish the efficacy of combined treatment with nepafenac and lubricant versus lubricant alone in improving epiphora and resolving punctal stenosis in Mexican adults.

DETAILED DESCRIPTION:
A two-month follow-up will be conducted. The study participants will be randomly assigned to two groups: the first group will receive treatment with nepafenac 0.1% ophthalmic suspension once daily and sodium carboxymethylcellulose 0.5% (lubricant) three times daily for eight weeks; the second group will receive treatment with placebo and lubricant only, administered three times daily for eight weeks. Initial evaluations will be conducted, followed by assessments at four and eight weeks to determine, through ophthalmological examination, the visibility of the lacrimal punctum using the Kashkouli scale, the assessment of epiphora according to the Munk scale, and the measurement of the external diameter and depth of the lacrimal punctum using OCT-SA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epiphora secondary to lacrimal punctum stenosis of allergic or idiopathic origin. Age ≥ 18 years

Exclusion Criteria:

* Previous eye surgery, including eyelid or lacrimal duct surgery. Allergy to nepafenac. Previous application of botulinum toxin to the eyelids, medical treatment received at least 3 months prior to the study, treatment discontinuation, failure to attend scheduled follow-up appointments and severe adverse reactions to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Lacrimal punctal estenosis | From enrollment to the end, each month of treatment until 8 weeks
  Lacrimal punctal stenosis measured by Optical Coherence Tomography and Kashkouli scale
Epiphora | From enrollment to the end, each month of treatment until 8 weeks
  Epiphora measured by Munk scale

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmología F.A.P. Conde de Valenciana, I.A.P., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2026 - December 2026

REFERENCES:
- [Result] Ceylanoglu KS, Sen EM. The effect of topical steroids and non-steroidal anti inflammatory drugs on epiphora of unknown cause: Optical coherence tomography study. Photodiagnosis Photodyn Ther. 2023 Mar;41:103234. doi: 10.1016/j.pdpdt.2022.103234. Epub 2022 Dec 5. PMID 36470407
- [Result] Assouline M, Renard G, Arne JL, David T, Lasmolles C, Malecaze F, Pouliquen YJ. A prospective randomized trial of topical soluble 0.1% indomethacin versus 0.1% diclofenac versus placebo for the control of pain following excimer laser photorefractive keratectomy. Ophthalmic Surg Lasers. 1998 May;29(5):365-74. PMID 9599360
- [Result] McGhee CN, Dean S, Danesh-Meyer H. Locally administered ocular corticosteroids: benefits and risks. Drug Saf. 2002;25(1):33-55. doi: 10.2165/00002018-200225010-00004. PMID 11820911
- [Result] Modi SS, Lehmann RP, Walters TR, Fong R, Christie WC, Roel L, Nethery D, Sager D, Tsorbatzoglou A, Philipson B, Traverso CE, Reiser H. Once-daily nepafenac ophthalmic suspension 0.3% to prevent and treat ocular inflammation and pain after cataract surgery: phase 3 study. J Cataract Refract Surg. 2014 Feb;40(2):203-11. doi: 10.1016/j.jcrs.2013.07.042. Epub 2013 Dec 15. PMID 24345529
- [Result] Teitel'baum IB. [Enterogenic phlegmon of the sigmoid]. Khirurgiia (Mosk). 1969 Jan;45(1):85-9. No abstract available. Russian. PMID 5768593
- [Result] Adolf J, Buttermann G, Theisinger W. [Effective prevention of thromboembolism with heparin and dihydroergotamine]. Med Klin. 1981 Jul 31;76(16):457-8. No abstract available. German. PMID 7266416
- [Result] Guidera AC, Luchs JI, Udell IJ. Keratitis, ulceration, and perforation associated with topical nonsteroidal anti-inflammatory drugs. Ophthalmology. 2001 May;108(5):936-44. doi: 10.1016/s0161-6420(00)00538-8. PMID 11320025
- [Result] Kessel L, Tendal B, Jorgensen KJ, Erngaard D, Flesner P, Andresen JL, Hjortdal J. Post-cataract prevention of inflammation and macular edema by steroid and nonsteroidal anti-inflammatory eye drops: a systematic review. Ophthalmology. 2014 Oct;121(10):1915-24. doi: 10.1016/j.ophtha.2014.04.035. Epub 2014 Jun 14. PMID 24935281
- [Result] Ambroziak AM, Szaflik J, Szaflik JP, Ambroziak M, Witkiewicz J, Skopinski P. Immunomodulation on the ocular surface: a review. Cent Eur J Immunol. 2016;41(2):195-208. doi: 10.5114/ceji.2016.60995. Epub 2016 Jul 15. PMID 27536206
- [Result] Moon I, Kang HG, Yeo A, Noh H, Kim HC, Song JS, Ji YW, Lee HK. Comparison of Ocular Surface Mucin Expression After Topical Ophthalmic Drug Administration in Dry Eye-Induced Mouse Model. J Ocul Pharmacol Ther. 2018 Nov;34(9):612-620. doi: 10.1089/jop.2018.0005. Epub 2018 Oct 16. PMID 30325678
- [Result] Holland EJ, Olsen TW, Ketcham JM, Florine C, Krachmer JH, Purcell JJ, Lam S, Tessler HH, Sugar J. Topical cyclosporin A in the treatment of anterior segment inflammatory disease. Cornea. 1993 Sep;12(5):413-9. doi: 10.1097/00003226-199309000-00008. PMID 8306663
- [Result] Nassief M, Lotfy NM. Topical cyclosporin A 0.05% eye drops for management of symptomatic acquired punctal stenosis: a prospective, controlled clinical study. Orbit. 2024 Apr;43(2):190-195. doi: 10.1080/01676830.2023.2232028. Epub 2023 Jul 18. PMID 37463348
- [Result] Vahdani K, Sian I, Giasin O, Makrygiannis G. Functional and anatomical outcomes of punctoplasty with Kelly punch. Eye (Lond). 2017 Nov;31(11):1628. doi: 10.1038/eye.2017.105. Epub 2017 Jun 2. No abstract available. PMID 28574492
- [Result] Wong ES, Li EY, Yuen HK. Long-term outcomes of punch punctoplasty with Kelly punch and review of literature. Eye (Lond). 2017 Apr;31(4):560-565. doi: 10.1038/eye.2016.271. Epub 2016 Dec 2. PMID 27911445
- [Result] Dolin SL, Hecht SD. The punctum pucker procedure for stenosis of the lacrimal punctum. Arch Ophthalmol. 1986 Jul;104(7):1086-7. doi: 10.1001/archopht.1986.01050190144055. PMID 3729781
- [Result] Hughes WL, Maris CS. A clip procedure for stenosis and eversion of the lacrimal punctum. Trans Am Acad Ophthalmol Otolaryngol. 1967;71(4):653-5
- [Result] Jones LT. The cure of epiphora due to canalicular disorders, trauma and surgical failures on the lacrimal passages. Trans Am Acad Ophthalmol Otolaryngol. 1962;66:506-24.
- [Result] Arlit F. Surgery of the lacrimal system. En: Graefe A, Saemisch T, editores. Handbook of the entire ophthalmology Leipzig, East Germany Publisher: Von Wilhelm Englemann. 1874
- [Result] Bowman W. Treatment method applicable to epiphora dependent on the outside reversal or obliteration of the lacrimal puncti. Ann Oculist. 1853;28:52-5
- [Result] Hussain RN, Kanani H, McMullan T. Use of mini-monoka stents for punctal/canalicular stenosis. Br J Ophthalmol. 2012 May;96(5):671-3. doi: 10.1136/bjophthalmol-2011-300670. Epub 2012 Jan 12. PMID 22241928
- [Result] Mathew RG, Olver JM. Mini-monoka made easy: a simple technique for mini-monoka insertion in acquired punctal stenosis. Ophthalmic Plast Reconstr Surg. 2011 Jul-Aug;27(4):293-4. doi: 10.1097/IOP.0b013e31820ccfaf. PMID 21386741
- [Result] Konuk O, Urgancioglu B, Unal M. Long-term success rate of perforated punctal plugs in the management of acquired punctal stenosis. Ophthalmic Plast Reconstr Surg. 2008 Sep-Oct;24(5):399-402. doi: 10.1097/IOP.0b013e318185a9ca. PMID 18806663
- [Result] Goldberg H, Priel A, Zloto O, Koval T, Varkel L, Ben Simon GJ. Kelly punch punctoplasty vs. simple punctal dilation, both with mini-monoka silicone stent intubation, for punctal stenosis related epiphora. Eye (Lond). 2021 Feb;35(2):532-535. doi: 10.1038/s41433-020-0891-3. Epub 2020 Apr 21. PMID 32317792
- [Result] Awny I, Mossa EAM, Bakheet TM, Mahmoud H, Mounir A. Changes of Lacrimal Puncta by Anterior Segment Optical Coherence Tomography after Topical Combined Antibiotic and Steroid Treatment in Cases of Inflammatory Punctual Stenosis. J Ophthalmol. 2022 Jan 24;2022:7988091. doi: 10.1155/2022/7988091. eCollection 2022. PMID 35111339
- [Result] Wawrzynski JR, Smith J, Sharma A, Saleh GM. Optical coherence tomography imaging of the proximal lacrimal system. Orbit. 2014 Dec;33(6):428-32. doi: 10.3109/01676830.2014.949793. Epub 2014 Sep 12. PMID 25215411
- [Result] Jiao H, Hill LJ, Downie LE, Chinnery HR. Anterior segment optical coherence tomography: its application in clinical practice and experimental models of disease. Clin Exp Optom. 2019 May;102(3):208-217. doi: 10.1111/cxo.12835. Epub 2018 Oct 1. PMID 30270476
- [Result] Munk PL, Lin DT, Morris DC. Epiphora: treatment by means of dacryocystoplasty with balloon dilation of the nasolacrimal drainage apparatus. Radiology. 1990 Dec;177(3):687-90. doi: 10.1148/radiology.177.3.2243969.
- [Result] Kashkouli MB, Nilforushan N, Nojomi N, Rezaee R. External lacrimal punctum grading: reliability and interobserver variation. Eur J Ophthalmol. 2008 Jul-Aug;18(4):507-11. doi: 10.1177/112067210801800401. PMID 18609466
- [Result] Offutt WN 4th, Cowen DE. Stenotic puncta: microsurgical punctoplasty. Ophthalmic Plast Reconstr Surg. 1993;9(3):201-5. doi: 10.1097/00002341-199309000-00006. PMID 8217962
- [Result] Kashkouli MB, Beigi B, Murthy R, Astbury N. Acquired external punctal stenosis: etiology and associated findings. Am J Ophthalmol. 2003 Dec;136(6):1079-84. doi: 10.1016/s0002-9394(03)00664-0. PMID 14644218
- [Result] Bukhari A. Prevalence of punctal stenosis among ophthalmology patients. Middle East Afr J Ophthalmol. 2009 Apr;16(2):85-7. doi: 10.4103/0974-9233.53867. PMID 20142967
- [Result] Kristan RW. Treatment of lacrimal punctal stenosis with a one-snip canaliculotomy and temporary punctal plugs. Arch Ophthalmol. 1988 Jul;106(7):878-9. doi: 10.1001/archopht.1988.01060140020006. No abstract available. PMID 3390040
- [Result] Esmaeli B, Valero V, Ahmadi MA, Booser D. Canalicular stenosis secondary to docetaxel (taxotere): a newly recognized side effect. Ophthalmology. 2001 May;108(5):994-5. doi: 10.1016/s0161-6420(00)00640-0. PMID 11320034
- [Result] Nassief M, Alduwailah OKM, Lotfy NM. Acquired symptomatic external punctal stenosis: a tertiary referral center study. Med Hypothesis Discov Innov Ophthalmol. 2021 May 31;10(1):18-23. doi: 10.51329/mehdiophthal1417. eCollection 2021 Spring. PMID 37641620
- [Result] Olver J. Colour Atlas of Lacrimal Surgery. Inglaterra: Butterworth-Heinemann; 2002
- [Result] Kakizaki H, Takahashi Y, Iwaki M, Nakano T, Asamoto K, Ikeda H, Goto E, Selva D, Leibovitch I. Punctal and canalicular anatomy: implications for canalicular occlusion in severe dry eye. Am J Ophthalmol. 2012 Feb;153(2):229-237.e1. doi: 10.1016/j.ajo.2011.07.010. Epub 2011 Oct 6. PMID 21982102
- [Result] Soiberman U, Kakizaki H, Selva D, Leibovitch I. Punctal stenosis: definition, diagnosis, and treatment. Clin Ophthalmol. 2012;6:1011-8. doi: 10.2147/OPTH.S31904. Epub 2012 Jul 3. PMID 22848141
- [Result] Awny I, Mossa EAM, Bakheet TM, Mahmoud H, Mounir A. Evaluation of Lacrimal Punctal Changes by Anterior Segment Optical Coherence Tomography after Punctal Dilation Versus Punctal Plug Insertion in Cases of Inflammatory Punctual Stenosis. J Ophthalmol. 2022 Oct 20;2022:7666323. doi: 10.1155/2022/7666323. eCollection 2022. PMID 36311352